CLINICAL TRIAL: NCT05807074
Title: The Impact of Tranexamic Acid in Reducing Hematoma and Seroma Formation in Reconstructive Post-oncologic Breast Surgery
Brief Title: Impact of Topical Tranexamic Acid in Breast Reconstruction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 228012; NCI-2023-02817 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-03-29; First posted 2023-04-10 (Actual); Results first posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast Reconstruction; Mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Tranexamic Acid; Sodium Chloride; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): Each participant will have one breast pocket exposed to TXA and the other to saline only prior to closure. During surgery and prior to wound closure, the wound surface will be moistened on one side with 20 cc of dilute TXA 25mg/ml solution, and the contralateral with 20cc of saline.
  Interventions: Drug: Tranexamic Acid; Other: Saline

INTERVENTIONS:
Drug: Tranexamic Acid — Applied intraoperatively
  Other Names: TXA; Lysteda
Other: Saline — Applied intraoperatively
  Other Names: Saline solution; Sodium Chloride 0.9%

SUMMARY:
Improvement in bleeding and bruising has been described by using both intravenous and topical off-label applications of Tranexamic Acid (TXA) in many surgical fields. This trial tests how well applying tranexamic acid (TXA) to the surface of the surgical site (topically) works to reduce post-operative bleeding (hematomas) and fluid collections (seromas) in women undergoing surgery to remove both breasts (bilateral mastectomy) immediately followed by surgery to rebuild the breast (reconstruction). The formation of hematomas and seromas, a common post-mastectomy complication, can interfere with breast reconstruction and increase the risk of infection and wound healing and can potentially delay cancer treatments. TXA is a synthetic molecule that pushes the body's clotting cascade toward clot formation to improve blood clotting. Applying TXA topically to the surgical site before closing the incision may prevent hematoma and seroma formation in post-mastectomy breast reconstruction patients.

Participants will be recruited from patients undergoing bilateral mastectomy at University of California, San Francisco.

DETAILED DESCRIPTION:
PRIMARY OUTCOMES:

I. To investigate whether topical tranexamic acid may impact rates of seroma, hematoma, severe bruising, and drain output in the post-mastectomy reconstructive population.

II. To evaluate the impact of TXA on seroma rates compared to control.

SECONDARY OUTCOMES:

I. To evaluate the impact of TXA on patient and provider rating of bruising, comparing the TXA side to the control side.

II. To evaluate the impact of TXA on total drain output in the first post operative day.

III. To evaluate the impact of TXA on total drain duration.

OUTLINE:

Participants will only be treated intra-operatively at the time of surgery with topical TXA to one breast pocket. Each participant will serve as own internal control, with one side receiving saline and the other TXA. Participants in this study will be assessed at their regularly scheduled visits up to one year post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed breast malignancy OR increased risk for breast cancer
2. Age >= 18 years
3. Scheduled to undergo bilateral mastectomy with plastic surgery closure or reconstruction
4. Ability to understand a written informed consent document, and the willingness to sign it
5. At least 4 weeks post-completion of chemotherapy or radiation therapy

Exclusion Criteria:

1. Any significant medical condition or laboratory abnormalities, which places the subject at unacceptable risk if she were to participate in the study
2. Any history of thromboembolic disease
3. Current anticoagulant use
4. Current use of chlorpromazine due to label contraindication
5. Current use of any prothrombotic medical products due to label contraindication
6. Documented or reported allergic reaction to tranexamic acid
7. Male participants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merisa Piper, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received the same intervention to the same breast pocket during bilateral mastectomy surgery before the study was closed prematurely to enrollment.
Units Other Than Participants: breast pocket
Groups:
- All Participants: Each participant received 20cc of dilute Tranexamic Acid (TXA) 25mg/ml solution in the pocket of the right breast during surgery and before wound closure and simultaneously administered 20 cubic centimeters (cc) of saline to the left breast pocket during surgery and before wound closure.
Period: Overall Study
Arm/Group | All Participants
Started | 23; 46 breast pocket (All participants were administered Tranexamic Acid (TXA) to the right breast)
Received TXA (Right Side) | 23; 23 breast pocket
Received Saline (Left Side) | 23; 23 breast pocket
Completed | 23; 46 breast pocket
Not Completed | 0; 0 breast pocket

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 23
Age, Customized [Count of Participants; unit: Participants]
  20-29 years old | 4
  30-39 years old | 4
  40-49 years old | 10
  50-59 years old | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Breast Pockets That Develop a Hematoma
Description: Presence of hematoma in the surgical area within a 30-day period from time of treatment application in the operating room will be reported.
Time Frame: Up to 1 month
Population: A total of 23 breast pockets received TXA, and a total of 23 breast pockets received saline for a total of 46 breast pockets
Measure: Number; unit: breast pocket
Units Other Than Participants: breast pockets
Arm/Group | All Participants
Number analyzed (Participants) | 23
Number analyzed (breast pockets) | 46
breast pocket
  TXA Breast Pocket: number analyzed (breast pockets) | 23
  TXA Breast Pocket | 0
  Saline Breast Pocket: number analyzed (breast pockets) | 23
  Saline Breast Pocket | 0

2. Primary Outcome: Number of Breast Pockets That Develop a Seroma
Description: Presence of seroma in the surgical area within 3-month period from time of treatment application in the operating room will be reported.
Time Frame: Up to 3 months
Population: as for outcome 1
Measure: Number; unit: breast pocket
Units Other Than Participants: breast pockets
Arm/Group | All Participants
Number analyzed (Participants) | 23
Number analyzed (breast pockets) | 46
breast pocket
  TXA Breast Pocket: number analyzed (breast pockets) | 23
  TXA Breast Pocket | 0
  Saline Breast Pocket: number analyzed (breast pockets) | 23
  Saline Breast Pocket | 0

3. Secondary Outcome: Number of Breast Pockets That Developed Ecchymosis
Description: Ecchymosis will be measured separately for the right and left breast pocket at each post operative visit and documented. The observer will be blinded to the laterality of TXA. Both participant and provider will be asked to rank which side, the right or left side, has worse bruising. The frequency of ecchymosis for the right and left side will be reported descriptively.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Number; unit: breast pockets
Units Other Than Participants: breast pockets
Arm/Group | All Participants
Number analyzed (Participants) | 23
Number analyzed (breast pockets) | 46
breast pockets
  TXA Breast Pocket: number analyzed (breast pockets) | 23
  TXA Breast Pocket | 0
  Saline Breast Pocket: number analyzed (breast pockets) | 23
  Saline Breast Pocket | 0

4. Secondary Outcome: Median Total Drain Output
Description: Total drain output over the life of the drain from drain placement in the operating room to discharge on post-operation day 1. Drains will be removed per standard practice at our institution which is when they have produced < 30 cubic centimeters (cc) per day for at least 3 days.
Time Frame: Approximately 1 month
Population: as for outcome 1
Measure: Median (Full Range); unit: cubic centimeter (cc) per day
Units Other Than Participants: breast pockets
Arm/Group | All Participants
Number analyzed (Participants) | 23
Number analyzed (breast pockets) | 46
cubic centimeter (cc) per day
  TXA Breast Pocket: number analyzed (breast pockets) | 23
  TXA Breast Pocket | 95 [35 to 293]
  Saline Breast Pocket: number analyzed (breast pockets) | 23
  Saline Breast Pocket | 90 [25 to 291]

5. Secondary Outcome: Median Total Drain Duration
Description: The median time of total drain duration from drain placement in the operating room to removal of the drain will be reported descriptively for the saline only and TXA treated breast.
Time Frame: Approximately 1 month
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Units Other Than Participants: breast pocket
Arm/Group | All Participants
Number analyzed (Participants) | 23
Number analyzed (breast pocket) | 46
days
  TXA Breast Pocket: number analyzed (breast pocket) | 23
  TXA Breast Pocket | 14 [8 to 32]
  Saline Breast Pocket: number analyzed (breast pocket) | 23
  Saline Breast Pocket | 14 [8 to 32]

6. Secondary Outcome: Number of Participants Requiring Reoperation After Completion of Bilateral Mastectomy
Description: The number of participants requiring an additional operation related to the bilateral mastectomy will be reported.
Time Frame: Up to 1 year
Population: It was pre-specified to assess reoperation in participants without regard to treatment, therefore data for TXA and Saline are combined in this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 23
Participants | 1

7. Secondary Outcome: Proportion of Participants With Reported Infection in Surgical Area Post-mastectomy
Description: The proportion of participants with demonstrated infection in surgical area related to the bilateral mastectomy will be reported.
Time Frame: Up to 1 year
Population: It was pre-specified to assess occurrence of post-surgical infection in participants regardless of breast pocket, therefore data for the TXA and Saline breast pockets are combined in this outcome measure
Measure: Number; unit: proportion of participants
Arm/Group | All Participants
Number analyzed (Participants) | 23
proportion of participants | 0.26

ADVERSE EVENTS:
Time Frame: Up to 1 year
Groups:
- Tranexamic Acid (TXA) (Right Side Breast Pocket); Saline (Left Side Breast Pocket): Each participant received 20cc of dilute Tranexamic Acid (TXA) 25mg/ml solution in the pocket of the right breast during surgery and before wound closure and simultaneously administered 20 cubic centimeters (cc) of saline to the left breast pocket during surgery and before wound closure.
Arm/Group | Tranexamic Acid (TXA) (Right Side Breast Pocket) | Saline (Left Side Breast Pocket)
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 3/23 | 3/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (TXA) (Right Side Breast Pocket) (N=23) | Saline (Left Side Breast Pocket) (N=23)
Breast Infection (Infections and infestations) | 3 (4) | 3 (4) — 3 participants (4 of 6 breasts) had infections in the TXA-treated breast, and 3 participants (4 of 6 breasts) had infections in the saline-treated breast

LIMITATIONS AND CAVEATS:
Study closed to enrollment earlier than expected due to slow accrual. As a result, all participants received the same intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT05807074/Prot_SAP_000.pdf